CLINICAL TRIAL: NCT06807931
Title: Impact of an Interactive Film-based Intervention on Resilience, Mental Wellbeing and Help-seeking Attitudes in Young People (14-18) At School Settings in North East of England: a Mixed-methods Cluster Randomised Controlled Feasibility Trial
Brief Title: Impact of an Interactive Film on Resilience, Wellbeing, and Help-Seeking in School-Aged Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sunderland (Other)
Collaborators: University of Huddersfield (Other); University of Cumbria (Unknown); Newcastle University (Other); North East and North Cumbria Child Health and Wellbeing Network (Unknown)
Responsible Party: Principal Investigator, Floor Christie-de Jong, Associate Professor in Public Health for Medicine, University of Sunderland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100471
Record Dates: First submitted 2025-01-17; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Mental Wellbeing; Resilience; Help-Seeking Behaviour
Keywords: Interactive film; Young people; School setting; Feasibility; Feasibility trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control condition (No Intervention): Participants in this condition received the standard Personal, Social, Health, and Economic (PSHE) Education curriculum provided by the school.
- Interactive Film (Experimental): Participants in this condition engaged in three class sessions wherein they watched the interactive film. The film was delivered both individually and to the whole class and featured decision points, and the viewer's choices influenced the storyline's progression.
  Interventions: Other: Interactive film
- Interactive Film Plus Support (Experimental): Participants in this condition watched the interactive film as in the previous condition. Additionally, they participated in facilitated discussions led by trained youth workers, focusing on the decisions made in the film and their consequences.
  Interventions: Other: Interactive film

INTERVENTIONS:
Other: Interactive film — An interactive film, co-produced with young people, that aims to provide young people with a virtual experience of making choices and facing consequences in various life scenarios. At key moments the action is paused and the user decides the outcome. The particular film series that was commissioned and included in the trial was 'Jessica's story', which focused on perinatal mental health, as well as many other public health issues relevant to young people, including mental wellbeing, domestic violence, and help-seeking behaviour.
  Arms: Interactive Film; Interactive Film Plus Support

SUMMARY:
The primary aim of this study is to assess the feasibility and acceptability of a randomised controlled trial of an interactive film intervention (commissioned through a North East and North Cumbria Child (NENC) Health & Wellbeing Network partnership and produced by Trylife), on building resilience, enhancing mental wellbeing and help-seeking attitudes for young people (14-18 years) in schools located in deprived areas of the North East and North Cumbria.

DETAILED DESCRIPTION:
Study Objectives:

* To conduct a three-arm feasibility trial to assess the feasibility of a brief interactive film intervention in school settings with randomisation at school level.
* To explore suitability of parameters of the trial, such as school recruitment, school randomisation, participant recruitment and retention, consent taking, data collection tools, feasibility and acceptability of the intervention, with a view of developing a large-scale trial, as primary outcome.
* To explore views and experiences of young people on acceptability and implementation of the trial and the film intervention through using a qualitative design.
* To gather preliminary data on the effectiveness of a brief interactive film intervention in school settings to enhance resilience, help-seeking attitudes and mental wellbeing in young people, as a secondary outcome.

Design Mixed-methods three arm feasibility cluster randomised controlled trial to assess the feasibility and acceptability of intervention delivery and study procedures, including the following key parameters: school recruitment and randomisation, sample size and participant recruitment and retention, consent taking, data collection tools, data analysis, intervention acceptability and delivery.

Setting Three schools across North East England and North Cumbria will be recruited, matched on size and socio-economic status, measured by percentage of children entitled to free meal.

School recruitment Schools will be recruited by telephoning and emailing head teachers at appropriate points of contact.

Randomisation Each of the three schools will be allocated at random (i.e. computer generated stratified randomisation), to one of the three intervention conditions: control condition, interactive film and interactive film plus support, matched according to the size of the school, socio-economic level, estimated by proportion of students receiving free school meals, and urban or rural location.

Participants Participants will be aged 14-18, years 10-12, at participating schools. Years 11 and 13 will not be targeted because of exam preparation, particularly in the light of COVID-19 disruption. Participants who receive parental consent as appropriate and who provide written informed consent/assent to taking part will be invited to complete baseline measures.

Study Intervention Interactive film

Follow-up Participants will be followed up at 3-months and 6-months.

Qualitative evaluation After the intervention participants will be invited to take part in a focus group (n=6, per school). Focus groups tend to be more comfortable for young people (29). The invitation will be on a separate form accompanying their survey documents. If participants are interested they will provide their contact details, which will be retained separately from the research data. The focus groups will explore young people's views on the trial procedures and the intervention. Interviews (n=6) will be conducted with head teachers and youth workers on acceptability of the trial and intervention.

Analysis Descriptive statistics will be used to provide estimations regarding recruitment, retention, intervention delivery and inform power-calculations for a large-scale trial.

Descriptive statistics will be used to report participants' scores on scales. Two-way ANOVA will be used for preliminary analysis to explore differences between groups, however instead of doing a formal hypothesis testing to prove effectiveness, a 95 % confidence interval will be presented to describe the range of effect.

Thematic content analysis will be used to capture recurring themes, commonalities and patterns in people's perspectives explored in focus groups and interviews.

ELIGIBILITY:
Inclusion Criteria:

* In selected Y10 or Y12 class (at start of study) at participating school

Exclusion Criteria:

* Lack of parental consent for Y10 students

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Willingness of schools to participate and be randomised | Qualitative data collection phase, month 20-23
  The qualitative assessment will be conducted through interviews with teachers and focus groups with students. They will be asked how they felt about randomisation and what, if any, challenges they encountered with this progression criterion.
Participant recruitment and retention | baseline, 3 and 6 month follow up
  Quantitative descriptive data, count number of participants at baseline, 3 and 6 month follow up
Suitability of data collection tools-Quantitative | Quantitative missing data, after 6 months Follow up
  Quantitative descriptive data, i.e. missing data
Suitability of data collection tools-qualitative perspectives | Qualitative data collection phase- month 20-23
  qualitative interviews and perspectives of participants on questionnaires, i.e. what did they think of the measures, length etc
Acceptability of the intervention | Qualitative data collection phase, study month 20-23
  qualitative exploration through focus groupd and interveiws-Was the intervention and its implementation acceptable to participants and stakeholders, including intervention components and delivery mode?
Feasibility of recruiting schools | Start intervention delivery - study month 6-
  Project monitoring data (descriptive data on number of schools and time of recruitment)
Feasibility of follow-up | After 6 months Follow up
  Descriptive quantitaive data-What proportion of participants could be followed up at 3 and 6 months?
Feasibility consent procedures | Qualitative data collection phase month 20-23
  Were consent procedures acceptable to participants? qualitative exploration through interviews and focus groups asking participants how they felt about consent procedures

SECONDARY OUTCOMES:
Mental wellbeing scale | Baseline, 3-months, 6-months
  Warwick Edinburgh Mental Wellbeing Scale (SWEMWBS), validated questionnaire. Scores raneg from 14-70 with higher scores indicating greater positive wellbeing
Resilience scale | Baseline, 3-months, 6-months
  Connor-Davidson Resilience Scale for young adults (10 items), validated questionnaire. Total scores range from 0-40, with higher scores indicating greater resilience
Help-seeking attitudes scale | Baseline, 3-months, 6-months
  The 10-item Attitudes Toward Seeking Professional Psychiatric Help Scale (ATSPPHS) tool, validated questionnaire Total range scores: 0-30, above 20 Reflect a positive attitude toward seeking professional psychological help. Below 10 Reflect a negative attitude or reluctance toward seeking professional psychological help.
  Mid range (10-20 Reflect ambivalence or mixed attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Floor Christie-de Jong, Principal Investigator — University of Sunderland
Locations (1):
- University of Sunderland, Sunderland, Sunderland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data can be shared upon reasonable request to the PI

REFERENCES:
- [Derived] Christie-de Jong F, Walker E, Corlett H, Hardarce C, Soulsby E, Arnott B, Franks K, Ling J, Stephenson J, Azevedo LB. A cluster randomised feasibility trial assessing an interactive film intervention to improve wellbeing of young people in school settings in the North of England. Pilot Feasibility Stud. 2025 Sep 2;11(1):117. doi: 10.1186/s40814-025-01699-1. PMID 40898276